CLINICAL TRIAL: NCT05543213
Title: The Effects of Action Observation Therapy (AOT) on Balance and Gait in Patients With Multiple Sclerosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Misagh Rahimi, Occupational Therapy expert, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 26181
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
Keywords: Action Observation; gait; Balance
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Videos of nature will be shown to them, and exercises similar to those in the intervention group will be practiced with them.
- Action Observation group (Active Comparator): In the intervention group, the same exercises related to balance and walking are practiced after watching videos of the exercises
  Interventions: Behavioral: Action Observation Therapy

INTERVENTIONS:
Behavioral: Action Observation Therapy — A video clip of a series of exercises is shown to the patients, then they practice them according to mirror neurons and observational learning.
  Arms: Action Observation group

SUMMARY:
Action observation therapy is a new method in rehabilitation that causes motor retraining by activating mirror neurons while watching the activity on the screen and then practicing them. We will use action observation therapy to improve balance and walking in MS patients.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an inflammatory disease of the brain and spinal cord caused by damage to myelin.

While the underlying cause of this disease is unknown, a significant relationship has been reported between a series of (CNS) neurons of the central nervous system, immune factors, genetics, and viruses. The primary complaint of MS patients is movement problems, particularly walking disorders, which greatly affect their quality of life, and its improvement is one of the main goals of rehabilitation. Action observation therapy is a new approach. It is used to treat neurological disorders such as cerebral palsy, Parkinson's disease, strokes, and multiple sclerosis.

In this method, a video of some purposeful movements and activities recorded by healthy people doing them is shown to the patient, then the person must try to imitate and perform those actions, which causes movement retraining and memory recall. Based on the studies conducted on the effectiveness of neurological treatment methods and proving the effectiveness of this method on other conditions, also considering the involvement of the nervous system in MS and the lack of related studies, we conducted this study with regard to To design a low cost, availability, and ease of use therapeutic method on balance and walking in patients with multiple sclerosis.

This study will be conducted on two groups of MS patients. after passing 30 minutes of usual rehabilitation by the blind therapist. One group will watch videos related to action observation exercises and then practice, and for the second group, a video of natural scenery will be shown for the same length of time, then they will practice exercises similar to the first group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic primary progressive, secondary progressive, relapsing-remitting MS
* EDSS (Extensive Disability Status Scale) Score between 3 and 6
* MMSE (Mini-mental state examination) test score> 24

Exclusion Criteria:

* Recurrence of MS during 3 months before intervention
* Pregnancy and lactation
* Having a psychiatric disorder or drug/alcohol abuse
* Changes in the symptoms of MS during the study period
* Inability to sit without torso support
* Inability to stand for at least 10 seconds with support
* Other neurological or orthopedic diseases of the lower extremities (musculoskeletal diseases, severe osteoarthritis, peripheral neuropathy, joint replacement)
* Cardiovascular diseases (recent myocardial infarction, heart failure, uncontrolled hypertension, orthostatic hypotension)
* participation in other clinical studies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 30 minutes
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Barthel Index | 25 minutes
  The Barthel Scale/Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.Time taken and physical assistance required to perform each item are used in determining the assigned value of each item. The Barthel Index measures the degree of assistance required by an individual on 10 items of mobility and self care ADL.
Functional Independence Measure (FIM) | 20 minutes
  The Functional Independence Measure (FIM) is an instrument that was developed as a measure of disability for a variety of populations and is not specific to any diagnosis. The FIM instrument
  Includes measures of independence for self-care, including sphincter control, transfers, locomotion, communication, and social cognition.
  Is an 18-item, seven-level, ordinal scale intended to be sensitive to changes over the course of a comprehensive inpatient medical rehabilitation program.
  Uses the level of assistance an individual needs to grade functional status from total independence to total assistance).
  The tool is used to assess a patient's level of disability as well as a change in patient status in response to rehabilitation or medical intervention.

SECONDARY OUTCOMES:
Fatigue Assessment Scale (FAS) | 10 minutes
  The Fatigue Assessment Scale (FAS) is a 10-item self-report scale evaluating symptoms of chronic fatigue. The FAS treats fatigue as a unidimensional construct and does not separate its measurement into different factors. However, in order to ensure that the scale evaluates all aspects of fatigue, it measures both physical and mental symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Taghi Karimi, PhD in OP, Study Chair — Full professor of orthotics and prosthetics
Locations (1):
- School of Rehabilitation Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
All data will be published in tables in the final article.